CLINICAL TRIAL: NCT07253311
Title: Evaluation of Rapid Diagnostic Device for the Detection of Candida Auris DiagRaMIE C AURIS
Brief Title: Evaluation of Rapid Diagnostic Device for the Detection of Candida Auris
Acronym: DiagRaMIE Caur
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: NG Biotech (Unknown); Commissariat A L'energie Atomique (Other Government)
Responsible Party: Sponsor
Other Study IDs: APHP 250168
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Candida Auris Infection; Candida Auris Colonization; Nosocomial Infections
Keywords: Candida auris; Diagnostic Tests; Routine; Immunochromatography; Microbiological Techniques; Sensitivity and Specificity; Microbial Drug Resistance, Fungal; Infection; Control
MeSH Terms: conditions — Candida auris infection; Cross Infection; Hypersensitivity; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: NG-TestⓇ C.auris kit — Evaluation of the performance of the rapid diagnostic test (RDT) for the detection of the Candida auris and comparision with MALDI-TOF result (reference test)

SUMMARY:
"Candida auris is an emerging fungus that can cause severe infections, particularly in hospitalized patients, and is often resistant to multiple antifungal treatments. Rapid and accurate detection of this pathogen is essential to control its spread in healthcare settings.

This study aims to evaluate the clinical performance of the NG-Test® Candida auris rapid diagnostic test (RDT), developed by CEA and NG Biotech. The test uses immunochromatography and can detect Candida auris in about 15 minutes. Its results will be compared to the reference method, MALDI-TOF, performed on colonies grown from routine patient samples.

Both retrospective (using stored isolates) and prospective (using new isolates) evaluations will be conducted. The study will measure the sensitivity and specificity of the test, and also include an assessment of its ease of use by laboratory staff. No additional samples will be collected from patients, and all testing will use de-identified isolates to ensure confidentiality."

DETAILED DESCRIPTION:
This monocentric, non-randomized diagnostic accuracy study aims to evaluate the NG-Test® Candida auris, a lateral flow immunoassay developed by CEA and NG Biotech, for the qualitative detection of Candida auris. Isolates will be obtained from patients with suspected infection or cutaneous colonization, grown on selective media from routine clinical samples, with no additional sampling. Test results will be compared with the reference method, MALDI-TOF. Approximately 224 isolates from infected patients and 330 isolates from colnized patients will be included, allowing precise estimation of sensitivity and specificity with 95% confidence intervals. Results from the rapid test, MALDI-TOF identifications, and pictures of the test cassettes will be entered into an electronic case report form under unique pseudonymized identifiers. Statistical analysis will include contingency tables, calculation of sensitivity, specificity, positive and negative predictive values, and likelihood ratios with 95% confidence intervals. Inter-observer agreement will be measured using Cohen's kappa coefficient. The study will be conducted over a six-month inclusion period in a single center, the Clinical Microbiology Laboratory of Attikon University Hospital in Athens. The validation of this rapid test is expected to provide a reliable tool to support infection control measures and limit the nosocomial spread of Candida auris.

ELIGIBILITY:
Inclusion Criteria:

From patients with suspected Candida auris infection:

- All isolates from the population that grow on the selective media: Sabouraud-dextrose (40g/L dextrose, 5.0g/L of peptic digest of animal tissue, 5.0 g/L of pancreatic digest of casein, 15.0 g/L of agar and final pH 5.6 ± 0.2) and CHROMagar™ Candida plus (manufactured by CHROMagar™, France). used in the hospital's routine diagnostic process.

From patients with suspected Candida auris cutaneous colonization:

- All isolates from the population that grow on the selective media: Salt-Sabouraud Dulcitol Broth (SSDB) with chloramphenicol and gentamicin (manufactured by S2 Media, United States), And the media used in the hospital's routine diagnostic process: Sabouraud Dextrose Liquid Medium containing NaCl 10%, chloramphenicol 50 mg/L.

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes hospitalized patients suspected of Candida auris infection or cutaneous colonization.
Sampling Method: Non-Probability Sample
Enrollment: 554 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
to evaluate the clinical performance of the NG-Test® Candida auris rapid diagnostic test (RDT), developed by CEA and NG Biotech, for detecting this pathogen using immunochromatography. | 1 day
  Sensitivity and specificity of the NG-Test® Candida auris rapid diagnostic test (RDT) will be assessed by comparison with the reference method (MALDI-TOF, Bruker) using colonies isolated prospectively from patients suspected of infection or colonization. The evaluation will also include a retrospective analysis using well-characterized isolates previously conserved by the microbiology department. Specificity will be assessed by testing a variety of non-Candida auris strains.

IPD SHARING:
Plan to Share IPD: No